CLINICAL TRIAL: NCT06964477
Title: A Randomized Controlled Trial of an Extended Reality-Based Occupational Therapy Intervention to Improve Leisure Participation in Inpatients With Persistent Mental Health Conditions
Brief Title: A Trial of Extended Reality Activities to Enhance Leisure Participation Among Inpatients With Persistent Mental Health Conditions
Acronym: XR-MHLP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chia-Hui Hung (Other)
Responsible Party: Sponsor-Investigator, Chia-Hui Hung, Associate Professor, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSTC 113-2410-H-040 -003 -MY3; CS1-24114 (Other: The Institutional Review Board Chung Shan Medical University Hospital)
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia and Related Disorders; Mental Disorders; Inpatients
Keywords: Leisure Activities; Virtual Reality Exposure Therapy; Augmented reality; Extend reality; Schizoaffective Disorder; Volition; Motivation; Emotional Regulation
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Psychotic Disorders; Self-Control; Emotional Regulation

STUDY DESIGN:
Masking Description: No blinding was implemented because the intervention involved observable differences between study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XR-Based Leisure Intervention (Experimental): Participants assigned to this arm will receive an extended reality (XR)-based leisure intervention that integrates both virtual reality (VR) and augmented reality (AR) technologies. The intervention is delivered once per week for six weeks. Each 40-minute session includes a 10-minute preparatory warm-up, a 20-minute immersive leisure experience using XR content, and a 10-minute structured feedback discussion. The XR experience is developed using the AR2VR platform and incorporates 360-degree panoramic video footage combined with interactive AR elements. The AR content is created using the MAKAR platform, a marker-based augmented reality development tool, enabling participants to interact with digital content through visual markers embedded in the physical or virtual environment. These AR features include interactive prompts, layered visuals, and context-based tasks designed to enhance engagement and therapeutic value.
  Interventions: Behavioral: XR-Based Leisure Intervention
- Standard Leisure Activities (Active Comparator): Participants assigned to this arm will engage in standard hospital-based leisure activities once per week for six weeks. Each session lasts approximately 40 minutes and includes a 10-minute warm-up, a 20-minute activity segment, and a 10-minute group discussion. Activities include therapeutic recreation commonly offered in psychiatric inpatient settings, such as drawing, music appreciation, newspaper reading, or light group exercises. The timing and structure of these sessions are designed to match those of the XR-based intervention group to ensure consistency in session duration and therapist involvement.
  Interventions: Behavioral: XR-Based Leisure Intervention

INTERVENTIONS:
Behavioral: XR-Based Leisure Intervention — The XR-based leisure intervention was developed based on occupational therapy principles and the therapeutic use of leisure to support engagement, volition, and emotional regulation in individuals with chronic mental illness. The intervention content was designed using the AR2VR platform and the MAKAR marker-based AR development system. Leisure scenarios were created by capturing real-world environments using 360-degree panoramic video and embedding interactive elements, such as contextual prompts, virtual objects, and multimedia cues, to enhance immersion and engagement.
  Sessions are guided by trained occupational therapists and follow a standardized protocol to ensure consistency. A simple cardboard VR viewer is used to reduce sensory overload and avoid adverse effects common with electronic head-mounted displays, such as dizziness or nausea. Activities target various leisure domains, including physical movement, creative expression, social activities, and cognitive play. Weekly con

SUMMARY:
The goal of this clinical trial is to evaluate the effects of an extended reality (XR)-enhanced occupational therapy leisure intervention on motivation, emotional engagement, and therapeutic participation among inpatients with chronic psychiatric conditions. The main questions it aims to answer are:

Can the XR intervention improve leisure motivation, leisure-related attitudes, and emotional coping strategies in long-term hospitalized individuals with mental illness?

Does the XR intervention promote improvements in psychological health, volition, and occupational performance?

Researchers will compare an XR-based leisure therapy group to a usual care group engaged in standard hospital leisure activities such as art, music, or reading. Participants will take part in weekly 40-minute sessions for 6 weeks. The XR group will use a custom-designed mobile VR program featuring immersive 360° leisure scenarios aligned with participants' interests and functional goals. Data collection includes standardized assessments (e.g., Interest Checklist, Volitional Questionnaire, COPM, PANSS) and semi-structured interviews to explore changes in motivation, coping, and perceived benefits.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effectiveness of an extended reality (XR)-based occupational therapy leisure intervention for inpatients with persistent mental health conditions. The study aims to improve patients' leisure motivation, leisure-related attitudes (including cognitive and behavioral engagement), emotional responses, and coping strategies through immersive therapeutic activities. It also examines the intervention's potential benefits for psychological well-being, volition, and occupational performance.

Participants are randomly assigned to either the experimental group or the control group. The experimental group receives an XR-enhanced leisure therapy program designed around three immersive features of extended reality: imagination, interaction, and immersion. The goal is to enhance the subjective quality of leisure experience and support the development of self-regulated leisure participation. Over a six-week period, participants in the intervention group will attend one 40-minute session per week, consisting of a 10-minute preparatory warm-up, a 20-minute immersive leisure experience utilizing virtual and augmented reality technologies, and a 10-minute structured feedback discussion.

The XR content is developed using the AR2VR application platform, integrating real-world 360-degree panoramic video footage of leisure environments. These environments are tailored to participants' interests, as identified using the Occupational Therapy Interest Checklist, and categorized according to eight types of leisure (e.g., physical activity, social interaction, hobbies, games, creative expression). The VR content includes embedded tasks, guided questions, audio-visual prompts, and simulated activities to stimulate engagement, cognition, and emotional regulation. To ensure safety and accessibility for individuals with chronic psychiatric conditions, a lightweight cardboard VR viewer is used instead of commercial electronic headsets. This approach minimizes the risk of sensory overstimulation, dizziness, or adverse events, which are more common in this population.

The control group participates in standard hospital leisure activities, such as newspaper reading, drawing, rhythmic movement, and basic group interactions. Both groups receive the intervention once weekly over six consecutive weeks.

Outcome evaluation includes both quantitative and qualitative data. Quantitative outcomes are assessed using validated tools:

The Occupational Therapy Interest Checklist measures leisure preferences and motivation.

The Volitional Questionnaire captures therapist-rated changes in volition during activity.

The Canadian Occupational Performance Measure (COPM) assesses participants' self-perceived competence and satisfaction in self-care, productivity, and leisure.

The Positive and Negative Syndrome Scale (PANSS) measures psychiatric symptom severity.

The Wellness Toolbox, a semi-structured interview tool, explores participants' emotional coping strategies before and after the intervention.

Qualitative data are collected through participant interviews and therapist observations and analyzed using grounded theory (open coding, axial coding, and selective coding). Quantitative data are analyzed using descriptive statistics and inferential statistics, including independent samples t-tests and repeated measures t-tests, to assess within- and between-group differences in outcome scores.

This study is expected to contribute new evidence regarding the therapeutic application of XR technologies in psychiatric settings and inform future models for integrating immersive digital tools into occupational therapy practice, particularly for enhancing engagement in meaningful leisure among individuals with long-term mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20 to 65 years
* Diagnosed with chronic schizophrenia or schizoaffective disorder (ICD-10 F20.x or F25.x)
* Hospitalized continuously for at least 6 months
* Clinically stable with no acute psychiatric symptoms
* Able to walk independently and communicate verbally
* Mini-Mental State Examination (MMSE) score ≥ 24

Exclusion Criteria:

* History of epilepsy, severe motion sickness, or other seizure-related conditions
* Significant visual or auditory impairments that may interfere with XR experience
* Physical conditions that limit participation in leisure activities
* Current diagnosis of substance abuse or major organic brain disorder
* Inability to distinguish between reality and virtual environments

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in Leisure Motivation Measured by the Occupational Therapy Interest Checklist | Baseline and after 6 weeks of intervention
  The Occupational Therapy Interest Checklist will be used to assess changes in leisure motivation, preferred activity domains, and engagement levels. Participants rate their interest in different activities before and after the 6-week intervention period.
Change in Occupational Performance and Satisfaction Measured by the Canadian Occupational Performance Measure | Baseline and after 6 weeks of intervention
  The Chinese version of the Canadian Occupational Performance Measure (COPM-C), originally developed by Law et al. and translated by Pan (2002), will be used to evaluate changes in self-perceived occupational performance and satisfaction. Participants identify up to five personally important occupational problems across three domains (self-care, productivity, and leisure) using a semi-structured interview. For each selected problem, participants rate their performance and satisfaction using a 10-point Likert scale. Higher scores indicate better performance or satisfaction. Final scores are calculated by averaging the performance and satisfaction ratings across the selected problems.
Change in Volition Observed Using the Volitional Questionnaire (VQ) | Weekly throughout the 6-week intervention period
  The Volitional Questionnaire (VQ), developed by de las Heras et al. based on the Model of Human Occupation, will be used to observe changes in participants' volition during occupational activity. The VQ includes 14 items categorized into three levels of volitional development: exploration, competence, and achievement. Trained occupational therapists observe participants during activity sessions and rate behaviors on a 4-point scale: passive, hesitant, involved, and spontaneous. Ratings reflect the degree of autonomy and internal motivation demonstrated during activity. Higher levels represent increased volitional expression and reduced therapist assistance.

SECONDARY OUTCOMES:
Change in Psychiatric Symptoms Measured by the Positive and Negative Syndrome Scale (PANSS) | Baseline and after 6 weeks of intervention
  The Positive and Negative Syndrome Scale (PANSS), developed by Kay, Opler, and Fiszbein (1987), will be used to evaluate changes in symptom severity among participants. The PANSS includes 30 items grouped into positive symptoms (7 items), negative symptoms (7 items), and general psychopathology (16 items), plus 3 additional items. Each item is scored from 1 (absent) to 7 (extreme), with total scores ranging from 30 to 231. Higher scores indicate more severe psychiatric symptoms. Severity categories are defined as mild (≤58), moderate (59-75), severe (76-95), and very severe (≥96).
Change in Emotional Coping Strategies Assessed Using the Wellness Toolbox Interview | Baseline and after 6 weeks of intervention
  The Wellness Toolbox is a semi-structured interview designed to explore participants' coping strategies for managing emotional distress and stress. It will be used to compare the number and types of self-reported strategies before and after the intervention. Participants will be asked to describe the strategies they typically use to regulate mood and handle stressful situations. Thematic and content analysis will be used to categorize qualitative changes, and the intervention's impact on emotional regulation and psychological well-being will be examined.

CONTACTS AND LOCATIONS:
Locations (1):
- Jing-Ho Hospital, Taichung, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No